CLINICAL TRIAL: NCT03024658
Title: Single Minute of Positive End Expiratory Pressure at the Time of Induction: Effect on Arterial Blood Gases and Hemodynamics in Morbidly Obese Patients Undergoing Laparoscopic Bariatric Surgery
Brief Title: Effect of Positive End Expiratory Pressure at the Time of Induction in Morbidly Obese Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sri Aurobindo Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Dr. Dipti Saxena, Associate Professor, Anaesthesiology, Sri Aurobindo Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Saims/IEC/14/02/35
Record Dates: First submitted 2017-01-06; First posted 2017-01-19 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2017-01

CONDITIONS: Morbid Obesity
Keywords: Pulmonary artery systolic pressure; Positive end expiratory pressure; morbidly obese; laparoscopic bariatric surgery
MeSH Terms: conditions — Obesity, Morbid | interventions — Positive-Pressure Respiration

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Zero PEEP (No Intervention): This group of patients did not receive any PEEP at the time of induction of general anesthesia (n= 30)
- PEEP- 10 cm of H2O (Experimental): This group comprised of patients who received a PEEP of 10 cm H2O at the time of induction of general anesthesia (n= 30)
  Interventions: Other: positive end expiratory pressure (PEEP)

INTERVENTIONS:
Other: positive end expiratory pressure (PEEP) — Positive end expiratory pressure was applied using anesthesia machine at the time of induction in the patients undergoing laparoscopic bariatric surgery
  Arms: PEEP- 10 cm of H2O

SUMMARY:
Background: Positive end expiratory pressure (PEEP) at the time of induction increases oxygenation by preventing lung atelectasis. However, PEEP may not prove beneficial in all cases. Factors affecting the action of PEEP have not been elucidated well and remain controversial. Pulmonary vasculature has direct bearing on the action of PEEP as has been proven in previous studies. Thus this study was planned to evaluate the action of PEEP on the basis of pulmonary artery systolic pressure (PASP) which is non invasive and easily measured by trans-thoracic echocardiography.

Methodology: This Randomized prospective study comprised of 70 morbidly obese patients, ASA grade II or III, aged 20-65 years with BMI > 40kg/m2, scheduled for elective laparoscopic bariatric surgery. Ten patients had to be excluded. Thus a total of 60 patients participated in the study. Thirty patients received no PEEP at the time of induction while other 30 patients were given a PEEP of 10cm of H2O. Serial ABG samples were taken pre operatively, at the time of intubation, 5 min after intubation and 10 min after intubation. Patients were then divided into four groups on the basis of PASP value of ≤ 30 mm Hg with and without PEEP or > 30 mm Hg

DETAILED DESCRIPTION:
This prospective study was conducted in the Department Of Anaesthesiology& Critical Care, Sri Aurobindo Institute of Medical Sciences & P.G. Institute and Mohak Hospitals, Indore, over a period of one year. Seventy morbidly obese patients, ASA grade II or III, aged 20-65 years with BMI > 40kg/m2, scheduled for elective laparoscopic bariatric surgery were selected and a written informed consent was obtained. All the recruited patients underwent 2D-trans-thoracic echocardiography and PASP was recorded. Echocardiography was performed by same cardiologist as this measurement is operator dependent. Patients who denied consent, those undergoing Emergency and/or open surgery and those requiring more than 2 attempts for intubation were excluded.

Arterial line was inserted pre operatively and ABG sample was taken and hemodynamic parameter recording done while the patient was breathing room air. Both groups were pre-oxygenated for 3 minutes with 100% Oxygen. Standard procedure was used for induction of anesthesia in all the patients. No premedication was given. All the patients were induced with i.v. Glycopyrolate (0.005-0.01 mg/kg), i.v. Fentanyl (2µg/kg) and i.v. Propofol. Once the patient became unresponsive to verbal commands, Succinylcholine was then administered in a dose of 1- 1.5 mg/ kg. Mechanical ventilation was started with 100% oxygen. A PEEP of 10 cm H2O was applied using four hand technique in Study group while the control group received no PEEP. After one minute endotracheal intubation was done. PEEP was continued in study group after intubation.

Arterial blood gas (ABG) analysis and hemodynamic parameters were recorded at following stages:

1. Just after inflation of cuff of endotracheal tube
2. 5 minutes post intubation
3. 10 minutes post intubation

Patients were then again divided into four groups on the basis of PASP:

Group 1: Patients with PASP ≤ 30 mmHg receiving no PEEP (n= 11) Group 2: PASP ≤ 30 mm Hg receiving PEEP of 10 cm H2O (n= 11) Group 3: PASP > 30 mm Hg receiving no PEEP (n= 19) Group 4: PASP > 30 mm Hg receiving PEEP of 10 cm H2O (n=19)

ELIGIBILITY:
Inclusion Criteria: Patients recruited were

* Anesthesia society of Anesthesiologist (ASA) physical status l, II or III,
* Aged 20-65 years
* BMI > 40kg/m2
* scheduled for elective laparoscopic bariatric surgery

Exclusion Criteria:

* Patients who denied consent
* Did not fulfill the inclusion criteria,
* patients undergoing Emergency and/or open surgery
* Patients requiring more than 2 attempts for intubation

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-05; Primary Completion 2016-06 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
effect of PEEP of 10 cm H2O on arterial blood gases and hemodynamic parameters, when applied at the time of induction | Arterial oxygenation (PaO2) in mm Hg recorded preoperatively and taken as baseline value
  Arterial oxygenation (PaO2) in mm Hg was recorded and compared between group receiving PEEP and group not receiving PEEP preoperatively just before taking the patient in operation theater
effect of PEEP of 10 cm H2O on arterial blood gases and hemodynamic parameters, when applied at the time of induction of general anesthesia | Arterial carbon di oxide (PaCO2) in mm Hg was recorded from ABG preoperatively and taken as baseline value
  Arterial carbon di oxide (PaCO2) values in mm Hg was recorded and compared between group receiving PEEP and group not receiving PEEP preoperatively just before taking the patient in operation theater
effect of PEEP of 10 cm H2O on arterial blood gases and hemodynamic parameters, when applied at the time of induction of general anesthesia | Pulse Rate (beats/ min) was recorded from ABG preoperatively and taken as baseline value
  Pulse Rate (beats/ min) was recorded and compared between group receiving PEEP and group not receiving PEEP preoperatively just before taking the patient in operation theater
effect of PEEP of 10 cm H2O on arterial blood gases and hemodynamic parameters, when applied at the time of induction of general anesthesia | Systolic BP in mm Hg was recorded from ABG preoperatively and taken as baseline value
  Systolic BP in mm Hg was recorded and compared between group receiving PEEP and group not receiving PEEP preoperatively just before taking the patient in operation theater
effect of PEEP of 10 cm H2O on arterial blood gases and hemodynamic parameters, when applied at the time of induction of general anesthesia | Diastolic BP in mm Hg was recorded from ABG preoperatively and taken as baseline value
  Diastolic BP in mm Hg was recorded and compared between group receiving PEEP and group not receiving PEEP preoperatively just before taking the patient in operation theater
effect of PEEP of 10 cm H2O on arterial blood gases and hemodynamic parameters, when applied at the time of induction | Arterial oxygenation (PaO2) in mm Hg was recorded just after the placement and cuff inflation of endotracheal tube
  Arterial oxygenation (PaO2) in mm Hg was recorded and compared between group receiving PEEP and group not receiving PEEP just after the placement and cuff inflation of endotracheal tube
effect of PEEP of 10 cm H2O on arterial blood gases and hemodynamic parameters, when applied at the time of induction | Arterial carbon di oxide (PaCO2) in mm Hg was recorded just after the placement and cuff inflation of endotracheal tube
  Arterial carbon di oxide (PaCO2) in mm Hg was recorded and compared between group receiving PEEP and group not receiving PEEP just after the placement and cuff inflation of endotracheal tube
effect of PEEP of 10 cm H2O on arterial blood gases and hemodynamic parameters, when applied at the time of induction | Pulse rate (beats/ min) was recorded just after the placement and cuff inflation of endotracheal tube
  Pulse rate (beats/ min) was recorded and compared between group receiving PEEP and group not receiving PEEP just after the placement and cuff inflation of endotracheal tube
effect of PEEP of 10 cm H2O on arterial blood gases and hemodynamic parameters, when applied at the time of induction | Systolic BP in mm Hg was recorded just after the placement and cuff inflation of endotracheal tube
  Systolic BP in mm Hg was recorded and compared between group receiving PEEP and group not receiving PEEP just after the placement and cuff inflation of endotracheal tube
effect of PEEP of 10 cm H2O on arterial blood gases and hemodynamic parameters, when applied at the time of induction | Diastolic BP in mm Hg was recorded just after the placement and cuff inflation of endotracheal tube
  Diastolic BP in mm Hg was recorded and compared between group receiving PEEP and group not receiving PEEP just after the placement and cuff inflation of endotracheal tube
effect of PEEP of 10 cm H2O on arterial blood gases and hemodynamic parameters, when applied at the time of induction | Arterial oxygenation (PaO2) in mm Hg was recorded five minutes post intubation
  Arterial oxygenation (PaO2) in mm Hg was recorded and compared between group receiving PEEP and group not receiving PEEP five minutes after intubation
effect of PEEP of 10 cm H2O on arterial blood gases and hemodynamic parameters, when applied at the time of induction | Arterial carbon di oxide (PaCO2) in mm Hg was recorded five minutes post intubation
  Arterial carbon di oxide (PaCO2) in mm Hg was recorded and compared between group receiving PEEP and group not receiving PEEP five minutes after intubation
effect of PEEP of 10 cm H2O on arterial blood gases and hemodynamic parameters, when applied at the time of induction | Pulse rate (beats/ min) was recorded five minutes post intubation
  Pulse rate (beats/ min) was recorded and compared between group receiving PEEP and group not receiving PEEP five minutes after intubation
effect of PEEP of 10 cm H2O on arterial blood gases and hemodynamic parameters, when applied at the time of induction | Systolic BP in mm Hg was recorded five minutes post intubation
  Systolic BP in mm Hg was recorded and compared between group receiving PEEP and group not receiving PEEP five minutes after intubation
effect of PEEP of 10 cm H2O on arterial blood gases and hemodynamic parameters, when applied at the time of induction | Diastolic BP in mm Hg was recorded five minutes post intubation
  Diastolic BP in mm Hg was recorded and compared between group receiving PEEP and group not receiving PEEP five minutes after intubation
effect of PEEP of 10 cm H2O on arterial blood gases and hemodynamic parameters, when applied at the time of induction | Arterial oxygenation (PaO2) in mm Hg was recorded ten minutes post intubation
  Arterial oxygenation (PaO2) in mm Hg was recorded and compared between group receiving PEEP and group not receiving PEEP ten minutes after intubation
effect of PEEP of 10 cm H2O on arterial blood gases and hemodynamic parameters, when applied at the time of induction | Arterial carbon di oxide (PaCO2) in mm Hg was recorded ten minutes post intubation
  Arterial carbon di oxide (PaCO2) in mm Hg was recorded and compared between group receiving PEEP and group not receiving PEEP ten minutes after intubation
effect of PEEP of 10 cm H2O on arterial blood gases and hemodynamic parameters, when applied at the time of induction | pulse Rate (beats/ min) was recorded ten minutes post intubation
  Pulse rate (beats/ min) was recorded and compared between group receiving PEEP and group not receiving PEEP ten minutes after intubation
effect of PEEP of 10 cm H2O on arterial blood gases and hemodynamic parameters, when applied at the time of induction | Systolic BP in mm Hg was recorded ten minutes post intubation
  Systolic BP in mm Hg was recorded and compared between group receiving PEEP and group not receiving PEEP ten minutes after intubation
effect of PEEP of 10 cm H2O on arterial blood gases and hemodynamic parameters, when applied at the time of induction | Diastolic BP in mm Hg was recorded ten minutes post intubation
  Diastolic BP in mm Hg was recorded and compared between group receiving PEEP and group not receiving PEEP ten minutes after intubation

SECONDARY OUTCOMES:
Effect of pulmonary artery systolic pressure (PASP) on the efficacy of PEEP as reflected by changes in ABG and hemodynamic parameters | ABG and hemodynamic parameters were recorded preoperatively and taken as baseline value
  Preoperative arterial oxygenation was compared of those patients who received PEEP and had PASP ≤ 30 mm Hg with those patients who did not receive PEEP and had PASP ≤ 30 mm Hg. Similarly the above parameter was compared in patients with PASP > 30 mm Hg receiving PEEP with those not receiving any PEEP
Effect of pulmonary artery systolic pressure (PASP) on the efficacy of PEEP as reflected by changes in ABG and hemodynamic parameters | ABG and hemodynamic parameters were recorded preoperatively and taken as baseline value
  Preoperative arterial carbon di oxide was compared of those patients who received PEEP and had PASP ≤ 30 mm Hg with those patients who did not receive PEEP and had PASP ≤ 30 mm Hg. Similarly the above parameter was compared in patients with PASP > 30 mm Hg receiving PEEP with those not receiving any PEEP
Effect of pulmonary artery systolic pressure (PASP) on the efficacy of PEEP as reflected by changes in ABG and hemodynamic parameters | ABG and hemodynamic parameters were recorded preoperatively and taken as baseline value
  Preoperative pulse rate was compared of those patients who received PEEP and had PASP ≤ 30 mm Hg with those patients who did not receive PEEP and had PASP ≤ 30 mm Hg. Similarly the above parameter was compared in patients with PASP > 30 mm Hg receiving PEEP with those not receiving any PEEP
Effect of pulmonary artery systolic pressure (PASP) on the efficacy of PEEP as reflected by changes in ABG and hemodynamic parameters | ABG and hemodynamic parameters were recorded preoperatively and taken as baseline value
  Systolic blood pressure was compared of those patients who received PEEP and had PASP ≤ 30 mm Hg with those patients who did not receive PEEP and had PASP ≤ 30 mm Hg. Similarly the above parameter was compared in patients with PASP > 30 mm Hg receiving PEEP with those not receiving any PEEP
Effect of pulmonary artery systolic pressure (PASP) on the efficacy of PEEP as reflected by changes in ABG and hemodynamic parameters | ABG and hemodynamic parameters were recorded preoperatively and taken as baseline value
  Diastolic blood pressure was compared of those patients who received PEEP and had PASP ≤ 30 mm Hg with those patients who did not receive PEEP and had PASP ≤ 30 mm Hg. Similarly the above parameter was compared in patients with PASP > 30 mm Hg receiving PEEP with those not receiving any PEEP
Effect of pulmonary artery systolic pressure (PASP) on the efficacy of PEEP as reflected by changes in ABG and hemodynamic parameters | ABG and hemodynamic parameters were recorded just after the placement and cuff inflation of endotracheal tube
  Arterial oxygenation recorded just after the placement and cuff inflation of endotracheal tube, was compared of those patients who received PEEP and had PASP ≤ 30 mm Hg with those patients who did not receive PEEP and had PASP ≤ 30 mm Hg. Similarly the above parameter was compared in patients with PASP > 30 mm Hg receiving PEEP with those not receiving any PEEP
Effect of pulmonary artery systolic pressure (PASP) on the efficacy of PEEP as reflected by changes in ABG and hemodynamic parameters | ABG and hemodynamic parameters were recorded just after the placement and cuff inflation of endotracheal tube
  Arterial carbon di oxide (mm Hg) recorded just after the placement and cuff inflation of endotracheal tube, was compared of those patients who received PEEP and had PASP ≤ 30 mm Hg with those patients who did not receive PEEP and had PASP ≤ 30 mm Hg. Similarly the above parameter was compared in patients with PASP > 30 mm Hg receiving PEEP with those not receiving any PEEP
Effect of pulmonary artery systolic pressure (PASP) on the efficacy of PEEP as reflected by changes in ABG and hemodynamic parameters | ABG and hemodynamic parameters were recorded just after the placement and cuff inflation of endotracheal tube
  Pulse rate (beats/ min) recorded just after the placement and cuff inflation of endotracheal tube, was compared of those patients who received PEEP and had PASP ≤ 30 mm Hg with those patients who did not receive PEEP and had PASP ≤ 30 mm Hg. Similarly the above parameters was compared in patients with PASP > 30 mm Hg receiving PEEP with those not receiving any PEEP
Effect of pulmonary artery systolic pressure (PASP) on the efficacy of PEEP as reflected by changes in ABG and hemodynamic parameters | ABG and hemodynamic parameters were recorded just after the placement and cuff inflation of endotracheal tube
  Systolic pressure(mm Hg) recorded just after the placement and cuff inflation of endotracheal tube, was compared of those patients who received PEEP and had PASP ≤ 30 mm Hg with those patients who did not receive PEEP and had PASP ≤ 30 mm Hg. Similarly the above parameter was compared in patients with PASP > 30 mm Hg receiving PEEP with those not receiving any PEEP
Effect of pulmonary artery systolic pressure (PASP) on the efficacy of PEEP as reflected by changes in ABG and hemodynamic parameters | ABG and hemodynamic parameters were recorded just after the placement and cuff inflation of endotracheal tube
  Diastolic blood pressure(mm Hg) recorded just after the placement and cuff inflation of endotracheal tube, was compared of those patients who received PEEP and had PASP ≤ 30 mm Hg with those patients who did not receive PEEP and had PASP ≤ 30 mm Hg. Similarly the above parameter was compared in patients with PASP > 30 mm Hg receiving PEEP with those not receiving any PEEP
Effect of pulmonary artery systolic pressure (PASP) on the efficacy of PEEP as reflected by changes in ABG and hemodynamic parameters | ABG and hemodynamic parameters were recorded five minutes post intubation
  Arterial oxygenation recorded five minutes after intubation, was compared of those patients who received PEEP and had PASP ≤ 30 mm Hg with those patients who did not receive PEEP and had PASP ≤ 30 mm Hg. Similarly the above parameter was compared in patients with PASP > 30 mm Hg receiving PEEP with those not receiving any PEEP
Effect of pulmonary artery systolic pressure (PASP) on the efficacy of PEEP as reflected by changes in ABG and hemodynamic parameters | ABG and hemodynamic parameters were recorded five minutes post intubation
  Arterial carbon di oxide (mm Hg) recorded five minutes after intubation, was compared of those patients who received PEEP and had PASP ≤ 30 mm Hg with those patients who did not receive PEEP and had PASP ≤ 30 mm Hg. Similarly the above parameter was compared in patients with PASP > 30 mm Hg receiving PEEP with those not receiving any PEEP
Effect of pulmonary artery systolic pressure (PASP) on the efficacy of PEEP as reflected by changes in ABG and hemodynamic parameters | ABG and hemodynamic parameters were recorded five minutes post intubation
  Pulse rate (beats/ min) recorded five minutes after intubation, was compared of those patients who received PEEP and had PASP ≤ 30 mm Hg with those patients who did not receive PEEP and had PASP ≤ 30 mm Hg. Similarly the above parameter was compared in patients with PASP > 30 mm Hg receiving PEEP with those not receiving any PEEP
Effect of pulmonary artery systolic pressure (PASP) on the efficacy of PEEP as reflected by changes in ABG and hemodynamic parameters | ABG and hemodynamic parameters were recorded five minutes post intubation
  Systolic pressure(mm Hg) recorded five minutes after intubation, was compared of those patients who received PEEP and had PASP ≤ 30 mm Hg with those patients who did not receive PEEP and had PASP ≤ 30 mm Hg. Similarly the above parameter was compared in patients with PASP > 30 mm Hg receiving PEEP with those not receiving any PEEP
Effect of pulmonary artery systolic pressure (PASP) on the efficacy of PEEP as reflected by changes in ABG and hemodynamic parameters | ABG and hemodynamic parameters were recorded five minutes post intubation
  Diastolic blood pressure(mm Hg) recorded five minutes after intubation, was compared of those patients who received PEEP and had PASP ≤ 30 mm Hg with those patients who did not receive PEEP and had PASP ≤ 30 mm Hg. Similarly the above parameter was compared in patients with PASP > 30 mm Hg receiving PEEP with those not receiving any PEEP
Effect of pulmonary artery systolic pressure (PASP) on the efficacy of PEEP as reflected by changes in ABG and hemodynamic parameters | ABG and hemodynamic parameters were recorded ten minutes post intubation
  Arterial oxygenation (mm Hg) recorded ten minutes after intubation, was compared of those patients who received PEEP and had PASP ≤ 30 mm Hg with those patients who did not receive PEEP and had PASP ≤ 30 mm Hg. Similarly the above parameter was compared in patients with PASP > 30 mm Hg receiving PEEP with those not receiving any PEEP
Effect of pulmonary artery systolic pressure (PASP) on the efficacy of PEEP as reflected by changes in ABG and hemodynamic parameters | ABG and hemodynamic parameters were recorded ten minutes post intubation
  Arterial carbon di oxide (mm Hg) recorded ten minutes after intubation, was compared of those patients who received PEEP and had PASP ≤ 30 mm Hg with those patients who did not receive PEEP and had PASP ≤ 30 mm Hg. Similarly the above parameter was compared in patients with PASP > 30 mm Hg receiving PEEP with those not receiving any PEEP
Effect of pulmonary artery systolic pressure (PASP) on the efficacy of PEEP as reflected by changes in ABG and hemodynamic parameters | ABG and hemodynamic parameters were recorded ten minutes post intubation
  Pulse rate (beats/ min) recorded ten minutes after intubation, was compared of those patients who received PEEP and had PASP ≤ 30 mm Hg with those patients who did not receive PEEP and had PASP ≤ 30 mm Hg. Similarly the above parameter was compared in patients with PASP > 30 mm Hg receiving PEEP with those not receiving any PEEP
Effect of pulmonary artery systolic pressure (PASP) on the efficacy of PEEP as reflected by changes in ABG and hemodynamic parameters | ABG and hemodynamic parameters were recorded ten minutes post intubation
  Systolic blood pressure (mm Hg) recorded ten minutes after intubation, was compared of those patients who received PEEP and had PASP ≤ 30 mm Hg with those patients who did not receive PEEP and had PASP ≤ 30 mm Hg. Similarly the above parameter was compared in patients with PASP > 30 mm Hg receiving PEEP with those not receiving any PEEP
Effect of pulmonary artery systolic pressure (PASP) on the efficacy of PEEP as reflected by changes in ABG and hemodynamic parameters | ABG and hemodynamic parameters were recorded ten minutes post intubation
  Diastolic blood pressure(mm Hg) recorded ten minutes after intubation, was compared of those patients who received PEEP and had PASP ≤ 30 mm Hg with those patients who did not receive PEEP and had PASP ≤ 30 mm Hg. Similarly the above parameter was compared in patients with PASP > 30 mm Hg receiving PEEP with those not receiving any PEEP

IPD SHARING:
Plan to Share IPD: Yes
data was recorded on a planned proforma. Masterchart was prepared on completion which is available for sharing.

REFERENCES:
- [Background] Reinius H, Jonsson L, Gustafsson S, Sundbom M, Duvernoy O, Pelosi P, Hedenstierna G, Freden F. Prevention of atelectasis in morbidly obese patients during general anesthesia and paralysis: a computerized tomography study. Anesthesiology. 2009 Nov;111(5):979-87. doi: 10.1097/ALN.0b013e3181b87edb. PMID 19809292
- [Result] Pelosi P, Croci M, Ravagnan I, Cerisara M, Vicardi P, Lissoni A, Gattinoni L. Respiratory system mechanics in sedated, paralyzed, morbidly obese patients. J Appl Physiol (1985). 1997 Mar;82(3):811-8. doi: 10.1152/jappl.1997.82.3.811. PMID 9074968
- [Result] Eichenberger A, Proietti S, Wicky S, Frascarolo P, Suter M, Spahn DR, Magnusson L. Morbid obesity and postoperative pulmonary atelectasis: an underestimated problem. Anesth Analg. 2002 Dec;95(6):1788-92, table of contents. doi: 10.1097/00000539-200212000-00060. PMID 12456460
- [Result] Coussa M, Proietti S, Schnyder P, Frascarolo P, Suter M, Spahn DR, Magnusson L. Prevention of atelectasis formation during the induction of general anesthesia in morbidly obese patients. Anesth Analg. 2004 May;98(5):1491-5, table of contents. doi: 10.1213/01.ane.0000111743.61132.99. PMID 15105237
- [Result] Almarakbi WA, Fawzi HM, Alhashemi JA. Effects of four intraoperative ventilatory strategies on respiratory compliance and gas exchange during laparoscopic gastric banding in obese patients. Br J Anaesth. 2009 Jun;102(6):862-8. doi: 10.1093/bja/aep084. Epub 2009 Apr 29. PMID 19403595
- [Result] Pelosi P, Goldner M, McKibben A, Adams A, Eccher G, Caironi P, Losappio S, Gattinoni L, Marini JJ. Recruitment and derecruitment during acute respiratory failure: an experimental study. Am J Respir Crit Care Med. 2001 Jul 1;164(1):122-30. doi: 10.1164/ajrccm.164.1.2007010. PMID 11435250
- [Result] Luecke T, Roth H, Joachim A, Herrmann P, Deventer B, Weisser G, Pelosi P, Quintel M. Effects of end-inspiratory and end-expiratory pressures on alveolar recruitment and derecruitment in saline-washout-induced lung injury -- a computed tomography study. Acta Anaesthesiol Scand. 2004 Jan;48(1):82-92. doi: 10.1111/j.1399-6576.2004.00265.x. PMID 14674978
- [Result] Gattinoni L, Pesenti A, Bombino M, Baglioni S, Rivolta M, Rossi F, Rossi G, Fumagalli R, Marcolin R, Mascheroni D, et al. Relationships between lung computed tomographic density, gas exchange, and PEEP in acute respiratory failure. Anesthesiology. 1988 Dec;69(6):824-32. doi: 10.1097/00000542-198812000-00005. PMID 3057937
- [Result] Maggiore SM, Jonson B, Richard JC, Jaber S, Lemaire F, Brochard L. Alveolar derecruitment at decremental positive end-expiratory pressure levels in acute lung injury: comparison with the lower inflection point, oxygenation, and compliance. Am J Respir Crit Care Med. 2001 Sep 1;164(5):795-801. doi: 10.1164/ajrccm.164.5.2006071. PMID 11549535
- [Result] Gattinoni L, Pesenti A, Baglioni S, Vitale G, Rivolta M, Pelosi P. Inflammatory pulmonary edema and positive end-expiratory pressure: correlations between imaging and physiologic studies. J Thorac Imaging. 1988 Jul;3(3):59-64. doi: 10.1097/00005382-198807000-00013. PMID 3292784
- [Result] Fougeres E, Teboul JL, Richard C, Osman D, Chemla D, Monnet X. Hemodynamic impact of a positive end-expiratory pressure setting in acute respiratory distress syndrome: importance of the volume status. Crit Care Med. 2010 Mar;38(3):802-7. doi: 10.1097/CCM.0b013e3181c587fd. PMID 19926983
- [Result] McQuillan BM, Picard MH, Leavitt M, Weyman AE. Clinical correlates and reference intervals for pulmonary artery systolic pressure among echocardiographically normal subjects. Circulation. 2001 Dec 4;104(23):2797-802. doi: 10.1161/hc4801.100076. PMID 11733397